CLINICAL TRIAL: NCT05871320
Title: Novel 99mTc-labeled Somatostatin Antaginosts in the Diagnostic Algotithm of Neuroendocrine Neoplasms - a Feasibility Study
Brief Title: Novel 99mTc-labeled Somatostatin Antaginosts in the Diagnostic Algotithm of Neuroendocrine Neoplasms
Acronym: TECANT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Collaborators: Medical University Innsbruck (Other); NCBJ Polatom: Narodowe Centrum Badań Jądrowych Polatom (Industry); University of Ljubljana (Other); University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Alicja Hubalewska-Dydejczyk, Professor, Jagiellonian University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TECANT; 2019-003379-20 (EudraCT Number)
Record Dates: First submitted 2023-02-07; First posted 2023-05-23 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Neuroendocrine Tumors
Keywords: Somatostatin receptors; neuroendocrine neoplasms; Positron emission tomography; Peptide Receptor Radionuclide Therapy; Single-photon emission computed tomography; SSTR2 antagonist; 99mTc; NEN tumour; Tc-99m-labeled SSTR2-Antagonist
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Intervention Model Description: Multi-center, Phase 0/I study, prospective single-arm, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [99mTc]Tc-TECANT1 (Experimental): The injection volume will be up to 5 mL over 20 seconds with an activity of 10 MBq/kg body weight (range between min. 500 and max. 800 MBq). To ensure application of the complete activity additionally 10 mL of 0.9% saline will be infused via the same system.
  Interventions: Drug: [99mTc]Tc-TECANT1

INTERVENTIONS:
Drug: [99mTc]Tc-TECANT1 — only one arm - the administration of [99mTC]-Tc-TECANT1 in all patients included

SUMMARY:
The main goal of the study is to expand cancer preclinical research results on the usefulness of SSTR2-Antagonist [99mTc]Tc-TECANT1 in clinical practice. Detection of NEN and monitoring of response to therapy is still challenging due to their cellular heterogeneity. Initial preclinical studies suggest that NEN imaging with the use of SSTR2-Antagonist may be advantageous in comparison to the widely used SSTR2-Agonists.

Recently, novel radiopharmaceuticals, based on SSTR2-Antagonists, were shown to provide superior SSTR2 visualisation than currently used agonists. The need for molecular imaging of NEN is expected to grow significantly in the near future due to their increasing incidence and prevalence. Although a persistent trend to shift the molecular imaging of NEN from conventional SPECT/CT gamma cameras to PET/CT has been observed in the last decade, labelling the compound with Tc-99m offers significant advantages by its extremely wide availability, low cost and low radiation exposure to patients. Effective and accessible molecular imaging methods as an integral part of personalised patient management are needed to optimise selection and follow-up of available therapeutic modalities. The Tc-99m-labeled SSTR2-Antagonist [99mTc]Tc-TECANT1 is expected to be an effective, widely available compound for quantitative assessment of SSTR2 NEN status, allowing a personalised therapeutic approach.

DETAILED DESCRIPTION:
Neuroendocrine neoplasms (NEN) are a heterogeneous group of malignancies that arise from various endocrine glands, endocrine cells within non-endocrine tissue and diffuse endocrine cells of the gastrointestinal, respiratory and genitourinary tract. Detection of NEN and monitoring of their response to therapy is challenging due to their varied location (often-unknown primary focus) and cellular heterogeneity. NEN exhibit a wide range of histological appearances and biological behaviors, and may all potentially behave in an aggressive manner, irrespective of the initial diagnosis. Consequently, the prediction of clinical outcomes in an individual patient is often difficult and inaccurate. According to some national registries, the incidence of NEN increased more than 6-fold and the prevalence more than 8-fold between 1973 and 2012, making NEN the second most prevalent diagnosis in gastrointestinal malignancies, thus representing a growing challenge. The rise in the incidence can be partly attributed to increased awareness of the disease and better detection methods. Diagnostic imaging is an integral part of the management of patients with NEN by localising the primary or recurrence site, determining the extent of the disease and evaluating response to therapy. Nuclear medicine with single-photon emission tomography (SPECT) and positron emission tomography (PET) is a branch of molecular imaging: in contrast to anatomical imaging, it depicts functional changes and biological characteristics of target tissues, providing a unique insight into the biology of malignant disease, and has established itself as an excellent tool in personalized medicine. The characteristic feature of NEN is an overexpression of somatostatin receptors (SSTR) on cell membranes. Molecular imaging techniques utilise the ability of SST analogues labelled with radioactive (single-photon or positron emitting) nuclides to bind to the SSTR. A combination of molecular and anatomical imaging (hybrid imaging, SPECT/CT and PET/CT) is currently the most sensitive approach to visualisation of SSTR-positive tumours. In NEN patients the prognosis depends on the grade and stage of the tumour. However, SSTR expression determines not only efficacy of staging using molecular imaging methods, but also efficacy of antiproliferative therapy with SST analogues both not radiolabelled ("cold") and labelled with a therapeutic radionuclide thus enabling Peptide Receptor Radionuclide Therapy (PRRT) as the main approach to personalised NEN patients' management. Traditionally, radiolabelled SST analogues were constructed aiming at their agonistic behaviour, based on their internalisation after SSTR activation and consequent retention within the tumour cells, believed to be crucial for efficient molecular imaging and therapy. Recently, it has been shown that novel molecular probes, SSTR antagonists, recognise more binding sites and hence improve diagnostic efficacy, especially when the density of SSTR is low. Accumulating preclinical and clinical data using both SPECT and PET tracers shows that high-affinity SSTR antagonists can provide better SSTR visualisation than agonists. Preclinical data and subsequent clinical evaluation demonstrated higher tumour uptake of an In-111-labelled antagonist [111In]In-DOTA-sst2-ANT ([111In]In-DOTA-BASS) compared to the agonist [111In]In-DTPA0-octreotide or [111In]In -DTPA0-octreotate, as well as superior tumour-to-background ratios. One of the first reports describing the SSTR2 antagonist LM3 indicates the high potential of gallium-68 (Ga-68) and copper-64 (Cu-64) radiolabelled LM3 in PET/CT. The authors demonstrated strong dependence of the affinity and pharmacokinetics of the SST-based radiolabelled antagonists on the chelator and radiometal, also confirmed using another SSTR antagonist, namely JR11. The Superiority of the SSTR antagonist was demonstrated in the Phase I/II clinical study using a positron emitter, [68Ga]Ga-NODAGA-JR11 and in a pilot study conducted with beta-emitting, therapeutic radionuclide (lutetium-177, Lu-177) labelled SSTR antagonist [177Lu]Lu-DOTA-JR11. As a result, research in the field is currently strongly focused on SSTR antagonists. Ga-68-labelled SST analogues have already established PET as a unique tool for personalising treatment of NEN. Nevertheless, single-photon emitting radiopharmaceuticals still represent the cornerstone of molecular imaging, particularly those based on Technetium-99m (Tc-99m). Its physical properties (half-life of 6 hours, optimal energy of 140 keV for imaging and lowest radiation exposure), widest on-site availability and cost-effectiveness are of major importance for routine clinical applications. Medical diagnostic imaging techniques using Tc-99m account for approximately 80% of all nuclear medicine procedures, representing 30-40 million examinations worldwide every year; even in developed countries, the number of gamma cameras in use exceeds by far the number of PET systems. Considering the above-mentioned characteristics Tc-99m is perfect for research with new radiotracers and is still recognised as the workhorse of diagnostic nuclear medicine. Quantifiable uptake of the radiopharmaceutical in target tissue using standardised methods and metrics such as standardised uptake value (SUV) is currently a unique feature of PET allowing highly personalized approaches to patient management and is part of clinical routine. It was shown also in NEN that the quantitative approach is able to adequately predict and evaluate the response to various treatments available, including "cold" and radiolabelled somatostatin analogues (PRRT). However, single-photon quantitative imaging has developed significantly and is also entering clinical routine. Identical quantitative metrics are becoming available with the use of SPECT/CT systems (SPECT SUV) with comparable accuracy and clinical applicability. The development of a quantitative SPECT imaging approach in NEN, in combination with improved, widely available radiopharmaceuticals, would therefore represent a highly significant improvement in management, tailored to the needs of each individual patient.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding and provision of signed and dated written informed consent by the patient or legally acceptable representative prior to any study-specific procedures.
2. Age ≥ 21 years
3. Male and female patients with cytologically/histologically confirmed NEN (G1 - G2) with SSTR positivity in molecular imaging (SPECT/PET - within 2 months before inclusion)
4. Karnofsky performance status ≥60%
5. Life expectancy of more than 6 months
6. Participating men must use a single barrier method for contraception for at least 6 months after completion of the trial starting at the day of application of [99mTc]Tc-TECANT1.
7. Women of childbearing age must use two highly effective methods of contraception during the trial and 6 months after application of investigational product if not in menopause or after hysterectomy.

The following contraceptive methods with a Pearl Index lower than 1% are regarded as highly effective:

* Oral hormonal contraception ("pill") (as far as its efficacy is not expected to be impaired during the trial, e.g. with IMPs that cause vomiting and diarrhoea, adequate safety cannot be assumed)
* Dermal hormonal contraception
* Vaginal hormonal contraception (NuvaRing®)
* Contraceptive plaster
* Long-acting injectable contraceptives
* Implants that release progesterone (Implanon®)
* Tubal ligation (female sterilisation)
* Double barrier methods This means that the following are not regarded as safe: condom plus spermicide, simple barrier methods (vaginal pessaries, condom, female condoms), copper spirals, the rhythm method, basal temperature method, and the withdrawal method (coitus interruptus).

The regulations for contraception are derived from Guideline ICH E8 Chapter 3.2.2.1 Selection of subjects together with ICH M3 note 4.

Exclusion Criteria:

1. Renal insufficiency with an eGFR <45 ml/min/1.73 m2 or intolerance to any constituents of intravenous CT-contrast agents
2. Higher than grade 2 hematotoxicity (CTC >2)
3. Co-existing malignancies (except non-melanoma skin carcinoma and uterine cervix carcinoma -in-situ unless without evidence of recurrence for 5 years)
4. Patients with concurrent illnesses/history of somatic/psychiatric disease that might preclude study completion or interfere with study results
5. Patients with bladder outflow obstruction or unmanageable urinary incontinence
6. Illness/clinically relevant trauma within 2 weeks before study entry
7. Pregnancy; breast-feeding; females planning to bear a child recently or with childbearing potential, unless a commonly accepted effective means of contraception is used
8. Prior administration of a radiopharmaceutical for SPECT-imaging within a period corresponding to 8 half-lives of the radionuclide used on such radiopharmaceutical.
9. Participation in any other investigational trial within 30 days of study entry with potential interactions regarding the study drugs or the underlying disease.
10. Known or expected hypersensitivity to somatostatin analogues or to any excipient of the study drug
11. History of somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study.
12. Clinically significant illness or clinically relevant trauma within 2 weeks before the administration of the investigational product.
13. Subjects with any kind of dependency on the investigator or is employed by the sponsor or investigator
14. Subjects held in an institution by legal or official order

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability assessment - incidence of Treatment-Emergent Adverse Events of iv administration of TECANT1 radiolabeled with 740±10% MBq of 99mTc | 14 days
  The number of patients with treatment-related adverse events as assessed by CTCAE v.5.0 (time frame: 2 weeks after administration)CTCAE v.5.0 (time frame: 2 weeks after administration)
Dosimetry assessment - effective dose absorbed in critical organs | 2 days
  Effective dose counted based on absorbed dose (energy deposited per unit mass) adjusted for radiation type and relative organ sensitivity measured in sievert (Sv)
Assessment of ionization radiation related to injection of TECANT1 | 2days
  Assessment of effective absorbed dose per injected activity [mSv/MBq] for critical organs (bone marrow, kidneys, bladder wall) and neoplastic lesions
Analysis of human pharmacokinetics of TECANT1 | 2 days
  1. Calculation of biological half-life of Tc-99m -SSTR2-Antagonist [99mTc]Tc-TECANT1 in blood (min) (based on time-activity curves)
  2. Assessment of the biological half-life of Tc-99m-SSTR2-Antagonist [99mTc]Tc-TECANT1 (min) in normal organs, tumour lesions (based on time-activity curves)

SECONDARY OUTCOMES:
Evaluation of [99mTc]Tc-TECANT01 uptake in tumour lesions. | 14 days
  Diagnostic accuracy assessed as the number of neoplastic lesions detected with [99mTc]Tc-TECANT1 in comparison to the number of lesions detected with ([68Ga]Ga-DOTA-TATE PET/CT)

CONTACTS AND LOCATIONS:
Overall Officials: Alicja Hubalewska-Dydejczyk, Prof., Principal Investigator — Endocrinology Clinic
Locations (3):
- Innsbruck Medical University Department of Nuclear Medicine, Innsbruck, Austria
- Department of Endocrinology, Jagiellonian University Medical College, Krakow, Poland
- University Medical Centre Ljubljana Department of Nuclear Medicine, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No